CLINICAL TRIAL: NCT00470912
Title: Photoprotective Effects of the RV 2457C Sunscreen Milk in Photoinduced Cutaneous Lupus Erythematosus
Brief Title: Sunscreen RV 2457C in Photoinduced CLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AMG 003
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: Cutaneous Lupus Erythematosus; Skin Lesion; Experimental Photoinduction; Protective Sunscreen
Keywords: cutaneous lupus erythemaosus; photoprotection; photoprovocation; Sunscreen RV 2547C
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sunscreen RV 2547C

SUMMARY:
Lupus erythematosus (LE) is characterized by a large clinical spectrum, and sunligt is a well established factor in the induction and exacerbation of this disease. In all subsets of LE, skin lesions occur preferentially in sun-exposed areas.

Previous studies have demonstrated that the lesions in LE patients reproduced in controlled experimental conditions. The initial reports suggested that the action spectrum for the LE was in the UVB range (290 to 320 nm), but more recent studies have demonstrated that UVA (320 to 400 nm) can contribute to the induction of LE skin lesions.

Antimalarial agents and topical steroids are the main treatments of chronic LE. The second line therapies include retinoids, sulfones, immunosuppressor agents, systemic corticosteroid and thalidomide. Moreover, patients are advised to avoid sun, to wear sunprotective clothing and to apply sunscreen.

The aim of this study was to assess the efficacy of a sunscreen milk with high protection factor against UV-B and UV-A, used exclusively, in the photoinduced LE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects
* Patient aged of 18 years or more
* Documented medical history of chronic cutaneous lupus erythematosus (lupus erythematosus tumidus, discoid lupus erythematosus, subacute lupus erythematosus) without any sign of systematic involvement
* patients who have a history of positive provocative phototestimg using a standardized protocol during a previous photobiologic exploration
* informed consent

Exclusion Criteria:

* Pregnant women, nursing mothers
* subjects with lupus erythematosus with systematic involvement
* subjects with a medical history of another photodermatosis
* subjects with sun erythema, residual pigmentation, dermatological lesion, abnormal skin pigmentation which might interfere with a study evaluation on test sides
* subjects who had sun solar simulator exposure on their backs within 12 weeks prior to enter to the study
* subjects with a known intolarance to one of the formula compounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2001-05; Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, MD, Principal Investigator — Heinrich-Heine University of Duesseldorf, Department of Dermatolgy
Locations (1):
- Heinrich Heine University of Duesseldorf, Depatment of Dermatoly, Düsseldorf, North Rhine-Westphalia, Germany